CLINICAL TRIAL: NCT02075008
Title: An Open-label, Multi-center, Extension Study to Evaluate the Long-term Safety of Subcutaneous 240mg QGE031 Given Every 4 Weeks for 52 Weeks in Allergic Asthma Patients Who Completed Study CQGE031B2201
Brief Title: Long-term Safety Study of QGE031 in Patients With Allergic Asthma Who Completed Study CQGE031B2201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated after core study CQGE031B2201 failed to meet the primary objective of demonstrating superiority for QGE031 versus placebo.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQGE031B2201E1; 2013-003683-31 (EudraCT Number)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: asthma; allergic asthma; QGE031; open-label; IgE; long-term safety
MeSH Terms: conditions — Asthma | interventions — ligelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QGE031 every 4 weeks (q4w) (Experimental): QGE031 240 mg subcutaneously q4w
  Interventions: Drug: QGE031

INTERVENTIONS:
Drug: QGE031 — QGE031 120 mg/mL solution for subcutaneous injection

SUMMARY:
This study planned to assess long-term safety of QGE031 during 12 months treatment in asthma patients who completed study CQGE031B2201.

DETAILED DESCRIPTION:
This study planned to assess long-term safety and tolerability of QGE031 administered every 4 weeks for an additional 12 months in patients with allergic asthma who previously completed study CQGE031B2201. The study was terminated early due to the efficacy results from an interim analysis of the Phase II study CQGE031B2201.

ELIGIBILITY:
Key Inclusion Criteria:

* forced Expiratory Volume in one second ( FEV1) >= 40% predicted
* patients who completed CQGE031B2201 study

Key Exclusion Criteria:

* life-threatening asthma attack, intubation, respiratory arrest during or after completion of CQGE031B2201 study
* new malignancy
* ongoing SAE from CQGE031B2201 that was assessed as related to study drug
* patient experienced platelets drop to < 75,000/uL
* patient experienced one unexpected grade 4 or two unexpected grade 3 hypersensitivity reactions
* patient is pregnant

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2016-03-22 (Actual); Study Completion 2016-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (76):
- United States (5):
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Fairfax, Virginia
- Argentina (9):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires F.D.
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Santa Fe
- Canada (3):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec
- Czechia (5):
  - Novartis Investigative Site, Trutnov, Czech Republic
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Břeclav
  - Novartis Investigative Site, Tábor
- Finland (2):
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (2):
  - Novartis Investigative Site, Le Kremlin
  - Novartis Investigative Site, Montpellier
- Germany (5):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Rüdersdorf
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Törökbálint
- Israel (4):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
- Italy (5):
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Verona, VR
- Novartis Investigative Site, Guadalajara, Jalisco, Mexico
- Poland (2):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lodz
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Romania (4):
  - Novartis Investigative Site, Bucharest, ROM
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
- Russia (5):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- Slovakia (6):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Prievidza
  - Novartis Investigative Site, Ružomberok
- Novartis Investigative Site, Berea, Durban, South Africa
- South Korea (6):
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Mersin
- United Kingdom (2):
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Southampton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, single arm study for participants who completed the core study CQGE031B2201 (NCT01716754).
Period: Overall Study
Arm/Group | QGE031 Every 4 Weeks (q4w)
Started | 270
Completed | 94
Not Completed | 176
Not completed — Technical problems | 1
Not completed — Pregnancy | 1
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1
Not completed — Death | 1
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 6
Not completed — Study terminated by Sponsor | 159

BASELINE CHARACTERISTICS:
Arm/Group | QGE031 Every 4 Weeks (q4w)
Number analyzed (Participants) | 270
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168
  Male | 102

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Participants With Non-serious Adverse Events (AEs), Serious AEs and Deaths as a Measure of Safety and Tolerability
Description: Safety was monitored throughout the study.
Time Frame: 52 weeks
Population: The safety set, which included all participants, was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | QGE031 Every 4 Weeks (q4w)
Number analyzed (Participants) | 270
Participants
  Non-serious AEs | 176
  Serious AEs | 19
  Deaths | 1

ADVERSE EVENTS:
Arm/Group | QGE031 Every 4 Weeks (q4w)
Serious Adverse Events (participants affected / at risk) | 19/270
Other Adverse Events (participants affected / at risk) | 130/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 Every 4 Weeks (q4w) (N=270)
Myocardial infarction (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Diverticulitis (Infections and infestations) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Vertebral artery thrombosis (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 5
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Varicose vein (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 Every 4 Weeks (q4w) (N=270)
Injection site reaction (General disorders) | 45
Bronchitis (Infections and infestations) | 20
Nasopharyngitis (Infections and infestations) | 33
Upper respiratory tract infection (Infections and infestations) | 17
Asthma (Respiratory, thoracic and mediastinal disorders) | 80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.